CLINICAL TRIAL: NCT03726268
Title: Optimizing Outpatient Anesthesia (OSPREy-Outpatient Surgery Pain Relief Enhancement)
Acronym: OSPREy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00089977; 1R01DA042985-01 (NIH)
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone; Fentanyl; Hydromorphone; Morphine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Short-stay, IV methadone (Active Comparator): Anticipated next-day discharge; intraoperative and post-operative IV methadone
  Interventions: Drug: Methadone
- Short-stay, IV short-acting opioids (Active Comparator): Anticipated next-day discharge; intraoperative and post-operative IV fentanyl, sufentanil, morphine, or hydromorphone at anesthesia provider discretion
  Interventions: Drug: Fentanyl; Drug: Hydromorphone; Drug: Morphine; Drug: Sufentanil
- Same-day, IV methadone (Active Comparator): Intraoperative and post-operative IV methadone
  Interventions: Drug: Methadone
- Same-day, IV short-acting opioids (Active Comparator): Intraoperative and post-operative IV fentanyl, sufentanil, morphine or hydromorphone at anesthesia provider discretion
  Interventions: Drug: Fentanyl; Drug: Hydromorphone; Drug: Morphine; Drug: Sufentanil

INTERVENTIONS:
Drug: Methadone — Dose is 0.15-0.3 mg/kg IV methadone HCl given intraoperatively and in the immediate post-operative period. Intraoperative methadone doses are 15 mg in "short-stay, anticipated next-day discharge" patients (10 mg if ≤55kg), and 10 mg in "same-day" surgery patients.
  Arms: Same-day, IV methadone; Short-stay, IV methadone
Drug: Fentanyl — Given per clinical provider discretion intraoperatively and in the immediate post-operative period (while patient remains in the post anesthesia care unit (PACU)).
  Arms: Same-day, IV short-acting opioids; Short-stay, IV short-acting opioids
Drug: Hydromorphone — Given per clinical provider discretion intraoperatively and in the immediate post-operative period (while patient remains in the post anesthesia care unit (PACU)).
  Arms: Same-day, IV short-acting opioids; Short-stay, IV short-acting opioids
Drug: Morphine — Given per clinical provider discretion intraoperatively and in the immediate post-operative period (while patient remains in the post anesthesia care unit (PACU)).
  Arms: Same-day, IV short-acting opioids; Short-stay, IV short-acting opioids
Drug: Sufentanil — Given per clinical provider discretion intraoperatively and in the immediate post-operative period (while patient remains in the post anesthesia care unit (PACU)).
  Arms: Same-day, IV short-acting opioids; Short-stay, IV short-acting opioids

SUMMARY:
The overall goal of this research is to improve perioperative pain treatment, decrease post-operative opioid consumption, diminish opioid related side effects, and reduce postop opioid prescribing (and hence opportunity for diversion, abuse, addiction, and fatal overdose).

DETAILED DESCRIPTION:
This protocol will test the innovative, paradigm-shifting hypothesis that anesthesia for outpatient surgery with long-duration opioids (methadone), compared with conventional short-duration opioids, achieves better analgesia, with similar or diminished side effects, may reduce development of chronic postsurgical pain, improves recovery, and importantly, decreases postoperative opioid consumption and could hence diminish take-home opioid prescribing and shrink the population reservoir of unused opioids available for diversion and misuse. Two cohorts will be studied, but analyzed separately. 1) Short-stay, anticipated next-day discharge surgery (compare short-duration vs long-duration opioid), 2) Same-day discharge surgery (compare short-duration vs long-duration opioid).

ELIGIBILITY:
Inclusion Criteria

* Age 18-65 years Undergoing general anesthesia and moderately painful ambulatory surgery with anticipated postop stay of < 24 hours
* Signed, written, informed consent

Exclusion Criteria

* History of liver or kidney disease.
* Females who are pregnant or nursing.
* Chronic opioid use (e.g. preoperative daily use of methadone, fentanyl transdermal patches, or ≥ 3 oxycodone pills)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 907 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Kharasch, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Short-stay, IV Methadone | Short-stay, IV Short-acting Opioids | Same-day, IV Methadone | Same-day, IV Short-acting Opioids
Started | 188 | 188 | 205 | 205
Completed | 175 | 175 | 190 | 194
Not Completed | 13 | 13 | 15 | 11
Not completed — Physician Decision | 2 | 8 | 6 | 3
Not completed — Withdrawal by Subject | 11 | 5 | 9 | 8

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Short-stay, IV Methadone | Short-stay, IV Short-acting Opioids | Same-day, IV Methadone | Same-day, IV Short-acting Opioids | Total
Number analyzed (Participants) | 175 | 175 | 190 | 194 | 734
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (13.4) | 41.6 (13.4) | 44.6 (12.3) | 43.6 (12.0) | 43.0 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 97 | 154 | 142 | 477
  Male | 91 | 78 | 36 | 52 | 257
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 7 | 8 | 25
  Not Hispanic or Latino | 161 | 164 | 171 | 173 | 669
  Unknown or Not Reported | 8 | 7 | 12 | 13 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 3 | 3 | 2 | 8
  Race: Asian | 2 | 4 | 1 | 5 | 12
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Race: Black or African American | 39 | 30 | 35 | 18 | 122
  Race: White | 124 | 131 | 140 | 164 | 559
  Race: More than one race | 2 | 0 | 4 | 1 | 7
  Race: Other | 2 | 2 | 4 | 1 | 9
  Race: Unknown or Not Reported | 6 | 5 | 3 | 3 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 175 | 175 | 190 | 194 | 734

OUTCOME MEASURES:

1. Primary Outcome: Total 30 Day Post-discharge Home Opioid Use (Number of Tablets)
Description: Based on home diary and hospital record. Number of opioid tablets from PACU discharge to postoperative day (POD) 30 for Same Day subjects, and number of opioid tablets from POD 1 to POD 30 for Short-Stay subjects.
Time Frame: Approximately 30 days
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Short-stay, IV Methadone | Short-stay, IV Short-acting Opioids | Same-day, IV Methadone | Same-day, IV Short-acting Opioids
Number analyzed (Participants) | 147 | 140 | 167 | 161
tablets | 10.00 (15.50) | 10.00 (11.60) | 6.18 (8.40) | 6.67 (10.40)
Statistical Analysis 1: Comparison: Short-stay, IV Methadone vs Short-stay, IV Short-acting Opioids; Test type: Other; p = 0.970, Negative binomial regression
Statistical Analysis 2: Comparison: Same-day, IV Methadone vs Same-day, IV Short-acting Opioids; Test type: Other; p = 0.631, Negative binomial regression

2. Secondary Outcome: Total Intraoperative Non-methadone Opioid Administration
Description: Based on hospital record.
Time Frame: Approximately 12 hours
Measure: Median (Inter-Quartile Range); unit: Milligram Morphine Equivalent (MME)
Arm/Group | Short-stay, IV Methadone | Short-stay, IV Short-acting Opioids | Same-day, IV Methadone | Same-day, IV Short-acting Opioids
Number analyzed (Participants) | 175 | 175 | 190 | 194
Milligram Morphine Equivalent (MME) | 0.0 [0.0 to 0.0] | 18.0 [14.0 to 23.0] | 0.0 [0.0 to 0.0] | 16.7 [12.7 to 24.0]
Statistical Analysis 1: Comparison: Short-stay, IV Methadone vs Short-stay, IV Short-acting Opioids; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Same-day, IV Methadone vs Same-day, IV Short-acting Opioids; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Total Post Anesthesia Care Unit (PACU) Opioid Administration
Description: Based on hospital record.
Time Frame: Approximately 2 hours
Measure: Median (Inter-Quartile Range); unit: Milligram Morphine Equivalent (MME)
Arm/Group | Short-stay, IV Methadone | Short-stay, IV Short-acting Opioids | Same-day, IV Methadone | Same-day, IV Short-acting Opioids
Number analyzed (Participants) | 175 | 175 | 190 | 194
Milligram Morphine Equivalent (MME) | 2.0 [0 to 4.0] | 3.0 [0.0 to 7.0] | 2.0 [0.0 to 4.0] | 2.5 [0.0 to 6.7]
Statistical Analysis 1: Comparison: Short-stay, IV Methadone vs Short-stay, IV Short-acting Opioids; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Same-day, IV Methadone vs Same-day, IV Short-acting Opioids; Test type: Other; p = 0.004, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Total Hospital Non-methadone Opioid Administration
Description: Based on hospital record.
Time Frame: Start of surgery to hospital discharge, up to 2 days
Measure: Median (Inter-Quartile Range); unit: Milligram Morphine Equivalent (MME)
Arm/Group | Short-stay, IV Methadone | Short-stay, IV Short-acting Opioids | Same-day, IV Methadone | Same-day, IV Short-acting Opioids
Number analyzed (Participants) | 175 | 175 | 190 | 194
Milligram Morphine Equivalent (MME) | 30 [0 to 80] | 128 [85 to 185] | 0 [0 to 15] | 68 [50 to 97]
Statistical Analysis 1: Comparison: Short-stay, IV Methadone vs Short-stay, IV Short-acting Opioids; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Same-day, IV Methadone vs Same-day, IV Short-acting Opioids; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Total 7-day Post-PACU Discharge Home Opioid Use
Description: Based on home diary and hospital record. Number of opioid tablets from PACU discharge to postoperative day (POD) 7 for Same Day subjects, and number of opioid tablets from POD 1 to POD 7 for Short-Stay subjects.
Time Frame: Up to 7 days post-PACU discharge
Population: Participants with data collected.
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Short-stay, IV Methadone | Short-stay, IV Short-acting Opioids | Same-day, IV Methadone | Same-day, IV Short-acting Opioids
Number analyzed (Participants) | 154 | 151 | 175 | 173
tablets | 6.50 (8.10) | 8.20 (8.70) | 4.96 (5.80) | 5.45 (7.20)
Statistical Analysis 1: Comparison: Short-stay, IV Methadone vs Short-stay, IV Short-acting Opioids; Test type: Other; p = 0.105, Negative binomial regression
Statistical Analysis 2: Comparison: Same-day, IV Methadone vs Same-day, IV Short-acting Opioids; Test type: Other; p = 0.531, Negative binomial regression

ADVERSE EVENTS:
Time Frame: Approximately 30 days
Arm/Group | Short-stay, IV Methadone | Short-stay, IV Short-acting Opioids | Same-day, IV Methadone | Same-day, IV Short-acting Opioids
All-Cause Mortality (participants affected / at risk) | 0/188 | 1/188 | 0/205 | 0/205
Serious Adverse Events (participants affected / at risk) | 6/188 | 6/188 | 10/205 | 11/205
Other Adverse Events (participants affected / at risk) | 21/188 | 17/188 | 29/205 | 16/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Short-stay, IV Methadone (N=188) | Short-stay, IV Short-acting Opioids (N=188) | Same-day, IV Methadone (N=205) | Same-day, IV Short-acting Opioids (N=205)
admission to behavioral facility (Psychiatric disorders) | 0 | 1 | 0 | 0
anastomotic leak (Gastrointestinal disorders) | 0 | 1 | 0 | 0
appendicitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
bladder spasms (Renal and urinary disorders) | 0 | 1 | 0 | 0
bleeding (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
bleeding ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
febrile neutropenia (Immune system disorders) | 1 | 0 | 0 | 0
fever (General disorders) | 1 | 0 | 1 | 0
colovesicular fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
seizures (Nervous system disorders) | 1 | 0 | 0 | 0
sepsis (Infections and infestations) | 0 | 1 | 0 | 0
urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Epistaxis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1
NSTEMI (Cardiac disorders) | 0 | 0 | 1 | 0
Post-operative Hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Vagal response to laryngoscopy (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1
cesarean delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
hemorrhagic cyst (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
pain (General disorders) | 0 | 0 | 1 | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
spontaneous labor (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Short-stay, IV Methadone (N=188) | Short-stay, IV Short-acting Opioids (N=188) | Same-day, IV Methadone (N=205) | Same-day, IV Short-acting Opioids (N=205)
COVID (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
DVT (Vascular disorders) | 1 | 1 | 1 | 0
abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0
abnormal ECG (Investigations) | 0 | 1 | 0 | 0
apnea (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 0 | 3
bladder spasms (Renal and urinary disorders) | 1 | 1 | 0 | 0
car accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
catheter placement (Surgical and medical procedures) | 0 | 1 | 0 | 0
elevated creatinine (Renal and urinary disorders) | 1 | 0 | 0 | 0
epistaxis (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
hives (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
hypertension (Cardiac disorders) | 0 | 1 | 0 | 0
hypotension (Cardiac disorders) | 2 | 0 | 1 | 1
hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
intraoperative decrease in compliance (Cardiac disorders) | 1 | 0 | 0 | 0
mouse bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
pain (General disorders) | 4 | 2 | 6 | 1
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
substance induced psychosis (Nervous system disorders) | 1 | 0 | 0 | 0
urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
intraoperative bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
RUE weakness (General disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
abscess (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
alcohol intoxication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
bladder defect (Renal and urinary disorders) | 0 | 0 | 0 | 1
bloody nasal discharge (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
convulsive-like movement (Nervous system disorders) | 0 | 0 | 1 | 0
diverticulitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
diverticulosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
eyelid swelling (Eye disorders) | 0 | 0 | 1 | 0
hand injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
headache (Nervous system disorders) | 0 | 0 | 1 | 0
heart palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
heart racing (Cardiac disorders) | 0 | 0 | 1 | 0
hematoma (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
leg cramps (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
levator spasms (Gastrointestinal disorders) | 0 | 0 | 1 | 0
mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0
nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
non-epileptic seizures (Nervous system disorders) | 0 | 0 | 0 | 1
pruritis (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
seizure (Nervous system disorders) | 0 | 0 | 1 | 0
seizure-like activity (Nervous system disorders) | 0 | 0 | 0 | 1
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
shoulder injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
somnolence (General disorders) | 0 | 0 | 1 | 0
tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
vaginal bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
ventilatory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
wound dressing (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT03726268/Prot_SAP_000.pdf